CLINICAL TRIAL: NCT04915755
Title: A Randomized Phase 3 Double-Blinded Study Comparing the Efficacy and Safety of Niraparib to Placebo in Participants With Either HER2-Negative BRCA-Mutated or Triple-Negative Breast Cancer With Molecular Disease Based on Presence of Circulating Tumor DNA After Definitive Therapy (ZEST)
Brief Title: Efficacy and Safety Comparison of Niraparib to Placebo in Participants With Human Epidermal Growth Factor 2 Negative (HER2-) Breast Cancer Susceptibility Gene Mutation (BRCAmut) or Triple-Negative Breast Cancer (TNBC) With Molecular Disease
Acronym: ZEST
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 213831; 2020-003973-23 (EudraCT Number)
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Neoplasms, Breast
Keywords: Niraparib; Breast cancer susceptibility gene; Human epidermal growth factor-2 negative (HER2); Breast cancer; Triple negative breast cancer (TNBC); Circulating tumor Deoxyribonucleic acid (ctDNA)
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — niraparib

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort1:Participants with tBRCAmut HER2-breast cancer(Independent of HR status,including HR+andTNBC) (Experimental): Eligible participants will receive either Niraparib or Placebo.
  Interventions: Drug: Niraparib; Drug: Placebo
- Cohort 2: Participants with tBRCAwt TNBC (Experimental): Eligible participants will receive either Niraparib or Placebo.
  Interventions: Drug: Niraparib; Drug: Placebo

INTERVENTIONS:
Drug: Niraparib — Niraparib will be administered.
Drug: Placebo — Matching placebo will be administered

SUMMARY:
This study will assess the efficacy and safety of Niraparib in participants with either tumor mutation in the BRCA gene (tBRCAmut) HER2- breast cancer (Independent of hormone receptor [HR] status, including HR positive [+] and TNBC) or tumor BRCA wild type (tBRCAwt) TNBC with molecular disease based on the presence of circulating tumor Deoxyribonucleic acid (ctDNA) following surgery or completion of adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Stage I to III breast cancer with surgical resection of the primary tumor that is confirmed to be either: TNBC, irrespective of BRCA status or HR+/HER2- breast cancer with a known and documented deleterious or suspected deleterious tBRCA mutation.
* Estrogen receptor (ER) and/or progesterone receptor (PgR) negativity is defined as immunohistochemistry (IHC) nuclear staining less than (<) 1 percentage (%), or by Allred scoring system where TNBC is defined to be 0 out of 8 or 2 out of 8, or staining in <1 % of cancer cells.
* Completed prior standard therapy for curative intent.
* Participants with HR+ breast cancer must be on a stable regimen of endocrine therapy.
* Detectable ctDNA as measured by central testing.
* An archival tumor tissue specimen of the primary tumor sufficient in quality and quantity for ctDNA assay design and tBRCA and Homologous recombination deficiency (HRD) testing is required.
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Prior treatment with a Poly Adenosine-diphosphate Ribose Polymerase (PARP) inhibitor.
* Current treatment with a Cyclin-dependent kinase (CDK)4/6 inhibitor or endocrine therapy other than anastrozole, letrozole, exemestane, and tamoxifen with or without ovarian suppression.
* Participants have any sign of metastasis or local recurrence after comprehensive assessment conducted per protocol.
* Participants have shown no definitive response to preoperative chemotherapy by pathologic, radiographic or clinical evaluation, in cases where preoperative chemotherapy was administered.
* Participants have inadequately treated or controlled hypertension.
* Participants have received live vaccine within 30 days of planned start of study randomization.
* Participants have a second primary malignancy.
* Exceptions are the following: (a) Adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, Ductal carcinoma in situ (DCIS) of the breast, Stage I Grade 1 endometrial carcinoma. (b) Other solid tumors and lymphomas (without bone marrow involvement) diagnosed >=5 years prior to randomization and treated with no evidence of disease recurrence and for whom no more than 1 line of chemotherapy was applied.
* Participant is pregnant, breastfeeding, or expecting to conceive children while receiving study treatment and/or for up to 180 days after the last dose of study treatment (except France).
* Participant is immunocompromised. Participants with splenectomy are allowed. Participants with known human immunodeficiency virus (HIV) are allowed if they meet protocol-defined criteria.
* Participants have a known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (163):
- United States (23):
  - GSK Investigational Site, Burbank, California
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Palo Alto, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Highlands Ranch, Colorado
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Skokie, Illinois
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Sioux Falls, South Dakota
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Everett, Washington
- Argentina (8):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Capital Federal
  - GSK Investigational Site, Cipoletti Rio Negro
  - GSK Investigational Site, Ciudad Autonoma Buenos Aires
  - GSK Investigational Site, Ciudad AutOnoma de Buenos Aire
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, Ciudad de Buenos Aires
  - GSK Investigational Site, Entre Ríos
- Australia (3):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Macquarie Park, New South Wales
  - GSK Investigational Site, North Sydney, New South Wales
- Austria (4):
  - GSK Investigational Site, Feldkirch
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Steyr
  - GSK Investigational Site, Vienna
- Belgium (4):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Charleroi
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
- Brazil (8):
  - GSK Investigational Site, Belo Horizonte
  - GSK Investigational Site, Florianópolis
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, Rio Grande
  - GSK Investigational Site, Salvador
  - GSK Investigational Site, São Paulo
  - GSK Investigational Site, Vitória
- Canada (4):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- Chile (2):
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Temuco
- Finland (2):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Turku
- France (9):
  - GSK Investigational Site, Avignon
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Saint-Cloud
- Germany (7):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Erlangen
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Mannheim
  - GSK Investigational Site, München
  - GSK Investigational Site, Ulm
- GSK Investigational Site, Debrecen, Hungary
- GSK Investigational Site, Dublin, Ireland
- Israel (6):
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Rehovot
  - GSK Investigational Site, Tel Aviv
- Italy (12):
  - GSK Investigational Site, Ancona
  - GSK Investigational Site, Bologna
  - GSK Investigational Site, Brindisi
  - GSK Investigational Site, Candiolo to
  - GSK Investigational Site, Catania
  - GSK Investigational Site, Genova
  - GSK Investigational Site, Meldola FC
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Monza
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Negrar Verona
  - GSK Investigational Site, Padua
- Japan (12):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo
- Mexico (3):
  - GSK Investigational Site, León
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Monterrey
- Netherlands (6):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Leeuwarden
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Zwolle
- Norway (2):
  - GSK Investigational Site, Drammen
  - GSK Investigational Site, Stavanger
- Poland (9):
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Rzeszów
  - GSK Investigational Site, Siedlce
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Portugal (2):
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Loures
- Romania (5):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Otopeni
  - GSK Investigational Site, Timișoara
- Russia (6):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Pushkin
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, StPetersburg
- South Africa (3):
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Port Elizabeth
  - GSK Investigational Site, Pretoria
- Spain (9):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Zaragoza
- GSK Investigational Site, Basel, Switzerland
- United Kingdom (11):
  - GSK Investigational Site, Bath
  - GSK Investigational Site, Brighton
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, Coventry
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London
  - GSK Investigational Site, Maidstone
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Sutton
  - GSK Investigational Site, Wigan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The results presented are based on the data cut-off date of 28 June 2024. Those participants still benefiting from study drug in the opinion of their treating physician continue to receive study drug in Post Analysis Continued Treatment (PACT) phase and their data will be reported after they stop receiving treatment as per protocol.
Groups:
- Niraparib: Participants with Either HER2-Negative BRCA-Mutated or Triple-Negative Breast Cancer received 200mg (two 100mg tablets) or 300 mg (three 100mg tablets) Niraparib tablet orally once daily depending on their body weight and platelet count, throughout each 28-day cycle starting on Cycle 1/Day 1 up to approximately 125 weeks.
- Placebo: Participants with Either HER2-Negative BRCA-Mutated or Triple-Negative Breast Cancer received Placebo tablet (two or three tablets) orally once a day depending on their body weight and platelet count, throughout each 28-day cycle starting on Cycle 1/Day 1 up to 64.7 weeks.
Period: Overall Study
Arm/Group | Niraparib | Placebo
Started (Intent-To-Treat Population included all participants randomized into the study.) | 18 | 22
Completed | 4 | 6
Not Completed | 14 | 16
Not completed — Physician Decision | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Ongoing for PACT | 3 | 2
Not completed — Other | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Niraparib | Placebo | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 58.1 (10.03) | 54.3 (14.22) | 56.0 (12.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race categories ('Asian' and 'Black or African American') are combined into 'All Other Races' category to maintain participant confidentiality and privacy.
  Participants
    White | 12 | 18 | 30
    Unknown | 0 | 1 | 1
    All other races | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Event (TEAEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose resulted in death, is life threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, is a congenital anomaly/birth defect, other situations and is associated with liver injury or impaired liver function. SAEs are subsets of AEs. TEAE is an event that emerged during treatment having been absent pretreatment or worsened relative to the pretreatment state. AESI is any AE (serious or nonserious) that is of scientific and medical concern specific to niraparib for which ongoing monitoring and rapid communication by the Investigator to the Sponsor is warranted. AEs were coded using the Medical Dictionary for Regulatory Activities (MedDRA) coding system.
Time Frame: Up to approximately 125 weeks
Population: Safety population included all randomized participants who received at least 1 dose of study treatment (niraparib or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib | Placebo
Number analyzed (Participants) | 18 | 22
Participants
  TEAEs | 18 | 17
  SAEs | 5 | 1
  AESIs | 0 | 0

2. Primary Outcome: Number of Participants With TEAEs Leading to Death
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAE is an event that emerged during treatment having been absent pretreatment or worsened relative to the pretreatment state.Number of participants with TEAEs leading to death were reported.
Time Frame: Up to approximately 125 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib | Placebo
Number analyzed (Participants) | 18 | 22
Participants | 0 | 0

3. Primary Outcome: Number of Participants With TEAEs Leading to Dose Modifications and Discontinuation of Study Treatment
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAE is an event that emerged during treatment having been absent pretreatment or worsened relative to the pretreatment state. Number of participants with TEAEs leading to dose modifications (reduction and interruption/delay) and permanent discontinuation of study treatment were reported.
Time Frame: Up to approximately 125 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib | Placebo
Number analyzed (Participants) | 18 | 22
Participants
  Dose reduction | 10 | 0
  Dose interruption/delay | 11 | 1
  Permanent discontinuation of study treatment | 0 | 0

4. Primary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: Number of participants with ECOG Performance Status was reported and was measured on 6-point grade scale 0: Fully active, able to carry on all pre-disease performance without restriction. Grade 1: Restricted in physically strenuous activity but ambulatory & able to carry out work of light or sedentary nature; Grade 2 - Ambulatory & capable of all self-care but unable to carry out any work activities. Up and about more than (>) 50% of waking hours; Grade 3 -Capable of only limited self-care, confined to bed or chair > 50% of waking hours; Grade 4 -Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; Grade 5 -Dead. Data is presented as baseline grade, best case on-therapy, and worst-case on-therapy for the available participants.
Time Frame: Up to approximately 125 weeks
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib | Placebo
Number analyzed (Participants) | 18 | 22
Participants
  Baseline, Grade 0 | 16 | 16
  Baseline, Grade 1 | 2 | 6
  Worst Case On-therapy, Grade 0: number analyzed (Participants) | 18 | 21
  Worst Case On-therapy, Grade 0 | 7 | 9
  Worst Case On-therapy, Grade 1: number analyzed (Participants) | 18 | 21
  Worst Case On-therapy, Grade 1 | 9 | 11
  Worst Case On-therapy, Grade 2: number analyzed (Participants) | 18 | 21
  Worst Case On-therapy, Grade 2 | 2 | 0
  Worst Case On-therapy, Grade 3: number analyzed (Participants) | 18 | 21
  Worst Case On-therapy, Grade 3 | 0 | 1
  Best Case On-therapy, Grade 0: number analyzed (Participants) | 18 | 21
  Best Case On-therapy, Grade 0 | 17 | 17
  Best Case On-therapy, Grade 1: number analyzed (Participants) | 18 | 21
  Best Case On-therapy, Grade 1 | 1 | 4

5. Primary Outcome: Number of Participants With Worst-Case Post-Baseline (WCPB) Hematology Results Relative to Baseline
Description: Blood samples were collected for the analysis of hematology parameters. The summaries of worst-case change from baseline with respect to normal range was analyzed for only those laboratory tests that were not gradable by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5. The number of participants with decreases to low from baseline, changes to normal or no changes from baseline, and increases to high values have been presented. Baseline is defined as the latest non-missing pre-dose value, including those from unscheduled visits.
Time Frame: Up to approximately 125 weeks
Population: Safety population. Only those participants with data available for specified parameter have been analyzed. Participants whose lab value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants are counted twice if the participant has values that changed 'To Low' and 'To High', so the percentages may not add to 100%.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib | Placebo
Number analyzed (Participants) | 18 | 22
Participants
  Basophils, To Low: number analyzed (Participants) | 16 | 20
  Basophils, To Low | 3 | 1
  Basophils, To Normal or No Change: number analyzed (Participants) | 16 | 20
  Basophils, To Normal or No Change | 12 | 19
  Basophils, To High: number analyzed (Participants) | 16 | 20
  Basophils, To High | 1 | 0
  Eosinophils, To Low: number analyzed (Participants) | 16 | 20
  Eosinophils, To Low | 4 | 3
  Eosinophils, To Normal or No Change: number analyzed (Participants) | 16 | 20
  Eosinophils, To Normal or No Change | 12 | 15
  Eosinophils, To High: number analyzed (Participants) | 16 | 20
  Eosinophils, To High | 0 | 2
  Erythrocyte Mean Corpuscular Volume (MCV), To Low | 1 | 1
  MCV, To Normal or No Change | 9 | 21
  MCV, To High | 9 | 0
  Hematocrit, To Low | 10 | 6
  Hematocrit, To Normal or No Change | 8 | 15
  Hematocrit, To High | 1 | 1
  Hemoglobin, To Low | 9 | 6
  Hemoglobin, To Normal or No Change | 9 | 16
  Hemoglobin, To High | 0 | 0
  Leukocytes, To Low | 13 | 2
  Leukocytes, To Normal or No Change | 3 | 19
  Leukocytes, To High | 4 | 1
  Lymphocytes, To Low | 9 | 1
  Lymphocytes, To Normal or No Change | 9 | 21
  Lymphocytes, To High | 0 | 0
  Monocytes, To Low: number analyzed (Participants) | 16 | 20
  Monocytes, To Low | 5 | 1
  Monocytes, To Normal or No Change: number analyzed (Participants) | 16 | 20
  Monocytes, To Normal or No Change | 10 | 17
  Monocytes, To High: number analyzed (Participants) | 16 | 20
  Monocytes, To High | 1 | 2
  Neutrophils, To Low | 9 | 6
  Neutrophils, To Normal or No Change | 8 | 14
  Neutrophils, To High | 3 | 2
  Platelets, To Low | 8 | 0
  Platelets, To Normal or No Change | 7 | 21
  Platelets, To High | 4 | 1

6. Primary Outcome: Number of Participants With Worst-Case Post-Baseline (WCPB) Clinical Chemistry Results Relative to Baseline
Description: Blood samples were collected for evaluation of clinical chemistry parameters. The summaries of worst case change from Baseline with respect to normal range have been presented for only those laboratory tests that are gradable by CTCAE v5.0. The number of participants with decreases to low, changes to normal or no changes from Baseline, and increases to high values have been presented. Baseline is defined as the latest non-missing pre-dose value, including those from unscheduled visits.
Time Frame: Up to approximately 125 weeks
Population: Safety population. Only those participants with data available for specified parameter have been analyzed.Participants whose lab value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants are counted twice if the participant has values that changed 'To Low' and 'To High', so the percentages may not add to 100%.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib | Placebo
Number analyzed (Participants) | 18 | 21
Participants
  Alanine aminotransferase (ALT), To Low | 0 | 1
  ALT, To Normal or No Change | 12 | 15
  ALT, To High | 6 | 5
  Albumin, To Low | 1 | 3
  Albumin, To Normal or No Change | 15 | 18
  Albumin, To High | 2 | 0
  Alkaline phosphatase (AP), To Low: number analyzed (Participants) | 18 | 20
  Alkaline phosphatase (AP), To Low | 1 | 0
  AP, To Normal or No Change: number analyzed (Participants) | 18 | 20
  AP, To Normal or No Change | 13 | 16
  AP, To High: number analyzed (Participants) | 18 | 20
  AP, To High | 4 | 4
  Amylase, To Low: number analyzed (Participants) | 8 | 7
  Amylase, To Low | 0 | 0
  Amylase, To Normal or No Change: number analyzed (Participants) | 8 | 7
  Amylase, To Normal or No Change | 8 | 7
  Amylase, To High: number analyzed (Participants) | 8 | 7
  Amylase, To High | 0 | 0
  Aspartate aminotransferase (AST), To Low | 0 | 0
  AST, To Normal or No Change | 12 | 18
  AST, To High | 6 | 3
  Bicarbonate, To Low: number analyzed (Participants) | 11 | 12
  Bicarbonate, To Low | 2 | 1
  Bicarbonate, To Normal or No Change: number analyzed (Participants) | 11 | 12
  Bicarbonate, To Normal or No Change | 5 | 9
  Bicarbonate, To High: number analyzed (Participants) | 11 | 12
  Bicarbonate, To High | 6 | 3
  Bilirubin, To Low: number analyzed (Participants) | 17 | 21
  Bilirubin, To Low | 2 | 3
  Bilirubin, To Normal or No Change: number analyzed (Participants) | 17 | 21
  Bilirubin, To Normal or No Change | 14 | 18
  Bilirubin, To High: number analyzed (Participants) | 17 | 21
  Bilirubin, To High | 2 | 0
  Calcium, To Low | 3 | 0
  Calcium, To Normal or No Change | 12 | 18
  Calcium, To High | 3 | 3
  Carbon Dioxide, To Low: number analyzed (Participants) | 4 | 4
  Carbon Dioxide, To Low | 0 | 0
  Carbon Dioxide, To Normal or No Change: number analyzed (Participants) | 4 | 4
  Carbon Dioxide, To Normal or No Change | 4 | 4
  Carbon Dioxide, To High: number analyzed (Participants) | 4 | 4
  Carbon Dioxide, To High | 0 | 0
  Chloride, To Low | 4 | 3
  Chloride, To Normal or No Change | 11 | 14
  Chloride, To High | 3 | 4
  Creatinine, To Low: number analyzed (Participants) | 18 | 20
  Creatinine, To Low | 1 | 1
  Creatinine, To Normal or No Change: number analyzed (Participants) | 18 | 20
  Creatinine, To Normal or No Change | 11 | 17
  Creatinine, To High: number analyzed (Participants) | 18 | 20
  Creatinine, To High | 6 | 2
  Direct Bilirubin, To Low: number analyzed (Participants) | 15 | 15
  Direct Bilirubin, To Low | 1 | 0
  Direct Bilirubin, To Normal or No Change: number analyzed (Participants) | 15 | 15
  Direct Bilirubin, To Normal or No Change | 12 | 13
  Direct Bilirubin, To High: number analyzed (Participants) | 15 | 15
  Direct Bilirubin, To High | 2 | 2
  Glucose, To Low | 1 | 2
  Glucose, To Normal or No Change | 11 | 13
  Glucose, To High | 7 | 6
  Lipase, To Low: number analyzed (Participants) | 3 | 4
  Lipase, To Low | 0 | 0
  Lipase, To Normal or No Change: number analyzed (Participants) | 3 | 4
  Lipase, To Normal or No Change | 3 | 4
  Lipase, To High: number analyzed (Participants) | 3 | 4
  Lipase, To High | 0 | 0
  Magnesium, To Low: number analyzed (Participants) | 9 | 8
  Magnesium, To Low | 1 | 1
  Magnesium, To Normal or No Change: number analyzed (Participants) | 9 | 8
  Magnesium, To Normal or No Change | 8 | 7
  Magnesium, To High: number analyzed (Participants) | 9 | 8
  Magnesium, To High | 0 | 0
  Phosphate, To Low: number analyzed (Participants) | 7 | 10
  Phosphate, To Low | 0 | 0
  Phosphate, To Normal or No Change: number analyzed (Participants) | 7 | 10
  Phosphate, To Normal or No Change | 5 | 10
  Phosphate, To High: number analyzed (Participants) | 7 | 10
  Phosphate, To High | 2 | 0
  Potassium, To Low | 2 | 2
  Potassium, To Normal or No Change | 13 | 16
  Potassium, To High | 3 | 3
  Protein, To Low: number analyzed (Participants) | 18 | 20
  Protein, To Low | 6 | 2
  Protein, To Normal or No Change: number analyzed (Participants) | 18 | 20
  Protein, To Normal or No Change | 11 | 17
  Protein, To High: number analyzed (Participants) | 18 | 20
  Protein, To High | 1 | 1
  Sodium, To Low | 3 | 1
  Sodium, To Normal or No Change | 14 | 19
  Sodium, To High | 1 | 1
  Urate, To Low: number analyzed (Participants) | 6 | 7
  Urate, To Low | 3 | 1
  Urate, To Normal or No Change: number analyzed (Participants) | 6 | 7
  Urate, To Normal or No Change | 2 | 6
  Urate, To High: number analyzed (Participants) | 6 | 7
  Urate, To High | 1 | 0
  Urea, To Low: number analyzed (Participants) | 15 | 15
  Urea, To Low | 0 | 1
  Urea, To Normal or No Change: number analyzed (Participants) | 15 | 15
  Urea, To Normal or No Change | 10 | 13
  Urea, To High: number analyzed (Participants) | 15 | 15
  Urea, To High | 5 | 1
  Urea Nitrogen, To Low: number analyzed (Participants) | 2 | 5
  Urea Nitrogen, To Low | 0 | 1
  Urea Nitrogen, To Normal or No Change: number analyzed (Participants) | 2 | 5
  Urea Nitrogen, To Normal or No Change | 2 | 3
  Urea Nitrogen, To High: number analyzed (Participants) | 2 | 5
  Urea Nitrogen, To High | 0 | 1

7. Primary Outcome: Number of Participants With Worst-Case Post-Baseline (WCPB) Vital Signs Results Relative to Baseline
Description: The abnormal vital sign ranges are: Pulse Rate (PR): Low [<60 beats per minute (bpm)], Normal (60 bpm to 100 bpm), High (>100 bpm); Temperature: Low (<35 degree Celsius (°C)), Normal (35 C and 38 C), High (>38 C); Systolic Blood Pressure (SBP): Low (<90 millimeter of mercury (mmHg)), Normal (>90 mmHg to <120 mmHg), High (>120 mmHg); Diastolic Blood Pressure (DBP): Low (<60 mmHg), Normal (60 mmHg to 79 mmHg), High (>80 mmHg). Participants were counted in the maximum worst case increase category that their value changes to (low, normal or high), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category.
Time Frame: Up to approximately 125 weeks
Population: Safety population. Only those participants with data available for specified parameter have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib | Placebo
Number analyzed (Participants) | 18 | 22
Participants
  DBP, To Low | 0 | 0
  DBP, To within Range or No Change | 13 | 22
  DBP, To High | 5 | 0
  PR, To Low | 1 | 4
  PR, To within Range or No Change | 9 | 16
  PR, To High | 8 | 2
  SBP, To Low | 0 | 0
  SBP, To within Range or No Change | 12 | 21
  SBP, To High | 6 | 1
  Temperature, To Low: number analyzed (Participants) | 18 | 21
  Temperature, To Low | 0 | 0
  Temperature, To within Range or No Change: number analyzed (Participants) | 18 | 21
  Temperature, To within Range or No Change | 18 | 21
  Temperature, To High: number analyzed (Participants) | 18 | 21
  Temperature, To High | 0 | 0

8. Primary Outcome: Number of Participants With Use of Concomitant Medications
Description: Number of participants who used concomitant medications is presented.
Time Frame: Up to approximately 125 weeks
Population: Intent-To-Treat Population included all participants randomized into the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib | Placebo
Number analyzed (Participants) | 18 | 22
Participants | 18 | 18

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected approximately 125 weeks. The results presented are based on data cut-off date 28 June 2024.
Description: All-cause mortality was reported for all enrolled participants. Safety population included all randomized participants who received at least 1 dose of study treatment (niraparib or placebo).
Arm/Group | Niraparib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 3/22
Serious Adverse Events (participants affected / at risk) | 5/18 | 1/22
Other Adverse Events (participants affected / at risk) | 18/18 | 17/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niraparib (N=18) | Placebo (N=22)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Subendocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niraparib (N=18) | Placebo (N=22)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 2 (4)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (3) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (2)
Dry eye (Eye disorders) | 1 (1) | 2 (2)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (11) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 6 (7)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Glossitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (7) | 6 (7)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 3 (3) | 4 (4)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 7 (8) | 7 (7)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 2 (2)
Mucosal inflammation (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (2) | 1 (2)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 3 (6) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (2) | 0 (0)
Cortisol decreased (Investigations) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (2) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (3) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Coital bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 6 (10) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT04915755/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT04915755/SAP_001.pdf